CLINICAL TRIAL: NCT03669055
Title: Radiological Study of the Hemodynamic Changes in the Aorta and Its Branches Before and After Endovascular Treatment of the Aortic Dissection
Brief Title: Hemodynamic Changes in the Aorta After Endovascular Treatment of the Aortic Dissection
Acronym: 4DAo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0361; 2018-A01742-53 (Other: n°ID-RCB)
Record Dates: First submitted 2018-07-30; First posted 2018-09-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Aortic Dissection
Keywords: aortic dissection; hemodynamic; 4D flow phase contrast MRI
MeSH Terms: conditions — Aortic Dissection | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-operative and post operative Magnetic Resonance Imaging (Experimental): Realization of an angio-MRI with 4D phase contrast sequence before and after the endovascular treatment of the aortic dissection
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Realization of a MRI before and after the endovascular treatment of the aortic dissection. Use of the 4D phase-contrast sequence during the MRI.

SUMMARY:
Aortic dissection (AD) is a serious pathology affecting one person for 300 000 habitants per year. In case of complicated AD on the descending aorta, it is necessary to perform an endovascular surgery in association with medical treatment. An endoprosthesis is implanted on the descending thoracic aorta in order to close the main intimal tear. This closure lead to an increase in the thoracic true lumen diameter, a decrease in the thoracic false lumen diameter, a better perfusion of the aortic branches. Furthermore, even in case of open surgical treatment of the ascending aorta it can be necessary to perform an endovascular treatment on the descending aorta, either to prevent and treat aneurysmal evolution or to treat patent malperfusion syndrome.

CT and Magnetic Resonance angiography, by the realization of an aortic morphologic evaluation, are the two key imaging exams in the DA. Nevertheless, CT can't provide aortic dynamic evaluation, contrary to MRI. This exam, thanks to the phase-contrast sequence can measure velocity and flow data in vessels, including aorta but also true and false lumen in the AD. Thus, by verifying the perfusion of the aortic true lumen and the aortic branches it is possible to perform an early evaluation of the endovascular treatment of the DA.

Actually, only one study has realized an aortic dynamic evaluation on the AD, unfortunately this study was limited to non-operated patients.

In order to assess the place of MRI in the AD, the ingestigation propose to determine if phase-contrast MRI is able to evaluate the impact of the endovascular treatment on the hemodynamic state of the aorta and its branches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an aortic dissection requiring endovascular treatment
* The endovascular treatment will be indicated according to the guidelines after medical, radiological and surgical multidisciplinary discussion in our hospital.
* Patients that have signed the informed consent form.
* Members of a social protection scheme.

Exclusion Criteria:

* Patients with an aortic dissection requiring an emergency intervention
* Patients with a contra-indication to endovascular treatment
* Contra-indication to MRI: claustrophobia, ferromagnetic materials: pacemaker, prosthetic heart valve, implantable cardioverter defibrillators, vascular clip
* Pregnancy
* Breastfeeding
* Dementia
* Patients under guardianship
* Patients with difficulty in understanding the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Comparative measurement of the flow in the aortic true lumen before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  The flows are measured in ml/s at several locations of the aortic true lumen. The flows are measured during the two MRI and compared with each other.

SECONDARY OUTCOMES:
Comparative measurement of the flow in the aortic false lumen before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  The flows are measured in ml/s at several locations of the aortic false lumen. The flows are measured during the two MRI and compared with each other.
Comparative measurement of the flow in the aortic branches before and after endovascular treatment of the aortic dissection | day 0 and day 16
  The flows are measured in ml/s in the celiac artery, the superior mesenteric artery, the inferior mesenteric artery, the right and left renal artery, the right and left primitive iliac artery.
  The flows are measured during the two MRI and compared with each other.
Comparative measurement of the number of intimal tear identified through 4D phase-contrast MRI relative to the number of intimal tear identified through Angio MRI before endovascular treatment of the aortic dissection | change from day 0 and day 16
  In the 4D phase-contrast MRI, an intimal tear is identified by a streamline going from the true lumen to the false lumen.
  In the Angio MRI, an intimal tear is identified by the visualization of the passage of the contrast agent from the true lumen to the false lumen.
Flow measurement through intimal tear with 4 Dimensions (4D) phase-contrast MRI before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  The intimal tears are identified thanks to the Angio MRI. The flows are measured during the two MRI and compared with each other.
Comparative measurement through 4D phase-contrast MRI of the shear forces before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  Shear forces are measured thanks to the 4D phase contrast MRI.
Comparative measurement through 4D phase-contrast MRI of parietal energy before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  Parietal energy is measured thanks to the 4D phase contrast MRI.
Comparative measurement through 4D phase-contrast MRI of the presence of helicoidal flow before and after endovascular treatment of the aortic dissection | change from day 0 and day 16
  The presence of a perpendicular flow to the main aortic flow is identified thanks to the 4D phase contrast MRI.
  The helicoidal flow is quantified by the degree of rotation between the beginning of the end of the cardiac cycle in millisecond.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No